CLINICAL TRIAL: NCT05313919
Title: Coronary Microcirculatory Disease and Inflammation in Patients With Chronic Coronary Syndrome and no Significant Coronary Artery Stenosis. MOSAIC-COR Study.
Brief Title: Coronary Microcirculatory Disease and Inflammation in Patients With Chronic Coronary Syndrome and no Significant Coronary Artery Stenosis
Acronym: MOSAIC-COR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bartlomiej Guzik (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor-Investigator, Bartlomiej Guzik, MD, PhD, John Paul II Hospital, Krakow
Organization: John Paul II Hospital, Krakow (Other)
Other Study IDs: 304/KBL/OIL2019; PL-2020-01 (Other Grant/Funding Number: Abbott)
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Coronary Artery Disease; Ischemia and No Obstructive Coronary Arteries; Ischemic Heart Disease; Microvascular Angina; Vasospastic Angina
Keywords: coronary artery disease; ischemia and no obstructive coronary arteries; ischemic heart disease; microvascular angina; vasospastic angina; coronary microvascular dysfunction; coronary microcirculation; endothelial dysfunction
MeSH Terms: conditions — Coronary Artery Disease; Ischemia; Myocardial Ischemia; Microvascular Angina; Angina Pectoris, Variant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1. Coronary microcirculatory disease
  Interventions: Diagnostic Test: Comprehensive functional diagnostics of coronary circulation
- 2. Epicardial vasospastic angina
  Interventions: Diagnostic Test: Comprehensive functional diagnostics of coronary circulation
- 3. Microvessel vasospastic angina
  Interventions: Diagnostic Test: Comprehensive functional diagnostics of coronary circulation
- 4. Non-cardiac disorder
  Interventions: Diagnostic Test: Comprehensive functional diagnostics of coronary circulation

INTERVENTIONS:
Diagnostic Test: Comprehensive functional diagnostics of coronary circulation — Comprehensive functional diagnostics of coronary circulation in patients with INOCA (ischemia and no obstructive coronary arteries) including:
  * echocardiography with assessment of diastolic function
  * flow-mediated dilation of brachial artery
  * coronary angiography
  * functional coronary assessment (RFR, FFR, IMR, CFR, dp/dt, Tau)
  * provocative test with acetylcholine (registration of symptoms, ECG and angiographic spasm)
  * laboratory tests (full blood count, serum creatinine level, eGFR, lipidogram, serum CRP/hsCRP level, serum NT-proBNP level)
  * serum level of inflammatory cytokines and chemokines

SUMMARY:
Patients with chronic coronary syndromes (CCS) diagnosed without significant lesions in invasive coronary angiography (ischemia non-obstructive coronary artery disease - INOCA) represent approximately 50% of all patients with CCS. Results of FAME study clearly showed that evaluation of coronary circulation should not be accomplished only with visual assessment in resting conditions. Current European Society of Cardiology Guidelines of diagnosis and treatment of CCS published in 2019 emphasize the necessity of performing complex coronary physiology assessment. Invasive physiological measurements and vasoreactivity provocative tests emerged as key tools to differentiate between vasospastic angina, microcirculatory angina, overlap of both conditions or non-cardiac disease. According to contemporary literature, identification of heterogeneity of patients with INOCA is crucial for determination of adequate treatment. An appropriate pharmacotherapy has a potential to improve outcomes including grade of angina, quality of life, exertional tolerance and most important - MACCE (major adverse cardiac and cardiovascular events) free survival. However, there is a lack of evidence on each of the subtypes of INOCA especially in those with signs and symptoms of vasospasm in provocative test but without visual spasm in epicardial vessels.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed chronic coronary syndrome CCS ≥ 2.
2. Evidence of myocardial ischemia (positive result of non-invasive stress test).
3. Informed consent.
4. Age at least 18 years.

Exclusion Criteria:

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic chronic coronary syndrome and no significant lesions in epicardial coronary arteries in angiography.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2020-07-24 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Cytokines (serum levels) | baseline
Diastolic Disfunction parameters in ECHO | baseline, 12- and 24-month follow-up

SECONDARY OUTCOMES:
MACCE occurrence | baseline, 12- and 24-month observation
Hospitalization any | baseline, 12- and 24-month observation
symptoms intensity and quality of life (questionnaires) | baseline, 12- and 24-month observation
FMD | baseline, 12- and 24-month observation

CONTACTS AND LOCATIONS:
Overall Officials: Bartłomiej Guzik, MD, PhD, Principal Investigator — John Paul II Hospital, Krakow, Poland; Jacek Legutko, MD, PhD, Professor, Study Director — John Paul II Hospital, Krakow, Poland
Locations (1):
- Department of Interventional Cardiology, John Paul II Hospital, Krakow, Poland, Institute Of Cardiology, Jagiellonian University Medical College, Krakow, Lesser Poland Voivodeship, Poland